| u |
|---------------|
| $\sigma$ |
| ~ |
| 900 |
| ب |
| - |
| _ |
| - 1 |
| $\simeq$ |
| 4 |
| C |
| _ |
| _ |
| 0 |
| 0 |
| 0 |
| ū |
| $\tilde{}$ |
| · |
| ~ |
| 1 |
| m |
| н |
| - 11 |
| Δ. |
| $\overline{}$ |
| ب |
| S |
| _ |
| ω |
| 4 |
| Ō |
| 059- |
| 0 |
| _ |
| ~ |
| m |
| _ |
| 7 |
| ~ |
| 0 |
| Œ |
| _ |

| Sponsor: | BIOTRONIK SE & Co KG |
|---|---|
| Study name / EAC code: | BIOSync CLS / BA103 |
| Version and date of the Statistical Analysis Plan: | 1-0, 19-FEB-2019 |
| Version and date of the underlying Clinical Investigation Plan: | 7-0, 20-JUN-2016 |

| Print Name & Title | Signature | Date of Signature (DD MMM YYYY) |
|---|---|---|
| Project Manager<br>Daniele Giacopelli | Davide Gree fall | 19-FEB-2019 |
| Scientist<br>Alessio Gargaro | e garage | 19 FB 2019 |
| Biostatistician<br>Alessio Gargaro | Slange | , 19 FEB 2019 |



# Page 2/14

# **Table of Contents**

| 1 | List of abbreviations | 3 |
|-----|----------------------------------------------|----|
| 2 | Introduction | 4 |
| 3.1 | Objectives | |
| 3.2 | Primary hypotheses | 4 |
| 3.3 | Secondary hypotheses | |
| 3 | Investigation plan | 5 |
| 4.2 | Inclusion criteria | 5 |
| 4.3 | Exclusion criteria | |
| 4.4 | Study procedures | |
| 4 | Determination of sample size | 6 |
| 5 | Database cleaning | 7 |
| 6 | Statistical methods | 7 |
| 7.1 | General methodology | |
| 7.2 | Handling of missing data | 7 |
| 7.3 | Baseline list variables | |
| 7.4 | Baseline data analysis | |
| 7.5 | Evaluation of study objectives | |
| 7.6 | Interim analysis | |
| 7.7 | Clinical Investigation Plan (CIP) deviations | |
| 7 | References | 14 |



# FOR-137- 059-B / SOP-137-060.020 / CRQ-15-00950

# 1 List of abbreviations

AV: Atrio-Ventricular BP: Blood Pressure

CDMS: Clinical Data Management System

CI: Confidence Interval

CIP: Clinical Investigation Plan CIR: Clinical Investigation Report CLS: Closed Loop Stimulation

CRO: Contract Research Organization CRT: Cardiac Resynchronization Therapy

CTL: Control group ECG: Electrocardiogram

eCRF: electronic Case Report Form ESC: European Society of Cardiology

HR: Hazard Ratio

ICD: Implantable Cardioverter Defibrillator IPG: Implantable Pulse Generator (pacemaker)

IRB/EC: Institutional Review Board/Ethics Committee

ITT: Intention to treat

LVEF: left ventricular ejection fraction

RCT: Randomized Clinical Trial SBP: Systolic Blood Pressure

TT: tilt table test



# 2 Introduction

The BIOSync CLS study is designed to test the hypothesis that DDD pacing with CLS stimulation is able to (completely or partially) prevent syncopal recurrences in patients with vaso-vagal syncope and documentated asysitolic pause at a pre-implant Tilt-Table test (TT).

## 3.1 Objectives

The study has the primary objective of comparing time to first syncopal recurrence between

- · active group (CLS): CLS in addition to DDD pacing mode; and
- control group (CTL): sensing only, ODO mode.

<u>Definition.</u> According to the 2018 ESC guidelines<sup>1</sup>, a syncopal recurrence is defined as a transient complete loss of consciousness characterized by rapid onset, short duration, and spontaneous complete recovery.

The Secondary endpoint will be the time to the first recurrence of pre-syncope or syncope, whichever comes first, compared between the study groups during follow-up

<u>Definition.</u> Pre-syncope is defined as any of the various signs and symptoms which are recognized by the patients as premonitory of imminent syncope but not followed by syncope.

# 3.2 Primary hypotheses

Null: the 2-year survival rate of syncopal recurrence in the treatment arm ( $S_{CLS}$ ) is equal to the 2-year survival rate of the control arm ( $S_{CTL}$ ), assuming an exponential distribution with proportional hazard rates.

 $H_0$ :  $S_{CLS}(t=2 \text{ years}) = S_{CTL}(t=2 \text{ years})$ 

Alternative: the 2-year survival rate of syncopal recurrence in the treatment arm is different from the 2-year survival rate of the control arm.

 $H_1$ :  $S_{CLS}(t=2 \text{ years}) \neq S_{CTL}(t=2 \text{ years})$ 

### 3.3 Secondary hypotheses

Null: the 2-year survival rate to the combined event of pre-syncope or syncope,  $\Sigma(t)$ , is equal in both study groups

 $H_0$ :  $\Sigma_{CLS}(t=2 \text{ years}) = \Sigma_{CTL}(t=2 \text{ years})$ 

Alternative: the 2-year survival rate to the combined event of pre-syncope or syncope is different in the two study groups.

 $H_1$ :  $\Sigma_{CLS}(t=2 \text{ years}) \neq \Sigma_{CTL}(t=2 \text{ years})$ 





# 3 Investigation plan

The study is a prospective, multi-center, double-blinded, randomized, intention-to-treat, placebo-controlled study.

Patients will be randomized to the active group or to placebo immediately after their enrolment and before any subsequent study-related procedure.

- Active group: before post-implant hospital discharge, IPG will programmed in a dualchamber DDD pacing mode with the CLS function ON.
- Control group: before post-implant hospital discharge, pacing will be programmed in the ODO mode.

Randomization ratio will be 1:1, therefore the randomization procedure will ensure that each individual patient will have (approximately) 50% chance to be assigned to the active group or to the control.

Patient selection adheres to the class IIb indication for cardiac pacing of the guidelines of the European Society of Cardiology<sup>1</sup>.

### 4.2 Inclusion criteria

Patients affected by clinical diagnosis of reflex (neurally-mediated) syncope who meet all the following criteria:

- age ≥40 years
- significant limitation of social and working life due to unpredictable frequent syncope recurrences, ≥2 of which within the last year.
- type 2B cardio-inhibitory response (VASIS classification) during TT performed according to the 'Italian protocol'.(7, 17)
- alternative therapies have failed or were not feasible.
- exclusion of other possible competitive causes of syncope.

### 4.3 Exclusion criteria

- Any classified indication to pacemaker different from reflex syncope with positive Tilt Test response
- Any classified indication implantable defibrillator (ICD), cardiac resynchronization therapy (CRT), according to current guidelines
- Any cardiac dysfunctions likely leading to loss of consciousness:
  - o overt heart failure;
  - o ejection fraction (LVEF) <40% (Echo-assessed within 3-month prior to study participation);
  - o myocardial infarction;
  - o diagnosis of hypertrophic or dilated cardiomyopathy;
  - o clinically significant valvular disease:
  - o sinus bradycardia <50 bpm or sinoatrial block;
  - o Mobitz I second degree atrioventricular block;
  - o Mobitz II second or third-degree atrioventricular block;
  - o bundle-branch block;





- o rapid paroxysmal supraventricular tachycardia or ventricular tachycardia;
- o pre-excited QRS complexes;
- o prolonged QT interval;
- o Brugada syndrome;
- o arrhythmogenic right ventricular cardiomyopathy;
- · Symptomatic orthostatic hypotension diagnosed by standing BP measurement;
- Nonsyncopal loss of consciousness (eg, epilepsy, psychiatric, metabolic, drop-attack, cerebral transient ischemic attack, intoxication, cataplexy).
- Symptomatic cardio-inhibitory carotid sinus hypersensitivity.

# 4.4 Study procedures

At enrolment, patients will receive anonymous syncope and pre-syncope assessment questionnaires to be self-administered upon each primary and secondary endpoint ever experienced and mailed (by ordinary mail) to an external CRO every 3 months after discharge b, using anonymous pre-paid and pre-addressed envelops.

Patients will be also visited in hospital at 12-, and 24-months. More frequent scheduled visits are optional and can be performed according to the site clinical practice. However, any scheduled or unscheduled in-hospital visit must be documented in the appropriate eCRF. Optionally, a 1-month  $(\pm 14 \text{ days})$  in-hospital visit may be performed to repeat the TT.

# 4 Determination of sample size

The study sample size calculation is based on the minimum relative difference in the 2-year incidence of syncopal recurrences as compared with placebo (pacemaker OFF).

The 2-year incidence of the primary endpoint in the control group will be assumed equal to the incidence observed in the control arm of the ISSUE 3 trial: <sup>2</sup> this was reported as high as 57%. The ISSUE 3 trial was considered as it selected a large population, had very similar inclusion/exclusion criteria, was recently published.

The BIOSync CLS study is designed to detect a 40% relative reduction of the 2-years incidence of syncopal recurrences (from 57% to 34%) with a statistical Type I and II errors of 0.05 (bilateral) and 0.20, respectively.

### Further assumptions:

- Exponential distribution of times to first recurrence
- Accrual time: 2 years
- Total study time: 4 years
- Randomization ratio: 1:1
- Loss incidence: 10% (both arms)

With these assumptions a sample size of 62 patients per study arm (124 in total) is required. This estimate must be further increased by 2%, due to the slight power loss induced by the interim analyses.

In summary, 128 subjects (64 per study arm) are necessary to reach the study primary objective with the required power.



The required number of primary endpoint events is 62, as calculated with the formula:

events = 
$$\frac{\left(z_{\alpha/2} + z_{\beta}\right)^{2}}{0.25 \log(HR)}$$

where  $z_{\alpha/2}$  and  $z_{\beta}$  are the standard normal percentiles ( $\alpha$ =0.05,  $\beta$ =0.20), HR is the expected hazard ratio. A HR of about 0.49 was calculated assuming an exponential model of the survival functions with proportional hazard rates.

# 5 Database cleaning

Data entered into the Clinical Data Management System (CDMS) is checked with programmed quality checks: input errors, discrepancies, missing data, and out-of-range values are resolved automatically (CDMS) or manually (clinical monitor, data manager) by means of data queries. The CDMS supports detailed tracking of the query process. Corrections to eCRF can only be done by the designated site personnel and need to be signed by the investigator. All changes are automatically recorded in the system's audit-trail.

### 6 Statistical methods

# 7.1 General methodology

Continuous variables will be summarized using tables of descriptive statistics: number of patients with recorded observations, mean, standard deviation, median, interquartile boundaries, minimum and maximum. Categorical variables will be summarized using counts and percentages. Descriptive statistics will be presented by randomization group.

Comparison of continuous parameters between two groups will be performed using T-test or Wilcoxon Man-Whitney U test, after testing for normality with the Shapiro-Wilk test. Categorical variables will be compared using the Chi-Square or Fisher exact test, as appropriate.

For the analysis of the primary and the secondary endpoint the Kaplan-Meier plots will be generated and the estimated survival functions of the study groups tested with the two- sided log-rank test. Dependence of survival on major baseline predictors will be evaluated with proportional hazard Cox models. Proportionality of hazards will be tested with the Schoenfeld Residuals test. Hazard ratios and relative 95% confidence intervals for each predictor will be calculated, respectively. Data will be censored at the date of last patient contact. The ITT principle will be applied.

All applicable statistical tests will be 2-sided and will be performed using a 5% significance level. All confidence intervals presented will be 95% and two-sided. Statistical calculations will be carried out by using STATA  $11.1 \, \text{@}$ , SAS  $9.3 \, \text{@}$  or R.

# 7.2 Handling of missing data

Missing or spurious data is not substituted; all data – as far as correctly measured – is analyzed. No method of imputation will be used for missing data.

In some cases, particular clinical data is excluded from analysis. The following reasons are possible:



FOR-137- 059-B / SOP-137-060.020 / CRQ-15-00950

- Data is not measured as described in the latest applicable version of the clinical investigation plan.
- Data is evaluated beyond the required follow-up schedule.
- Patient has to be excluded because she/he does not fulfill the exclusion/inclusion criteria.
- Patient requires that all recorded data has to be deleted.
- There is evidence of incomplete or incorrect patient consent process.

### **Baseline list variables** 7.3

The following table reports the description of relevant baseline variables.

| Variable name | List of values | Unit of measure | Description |
|---|---|---|---|
| rd_display | 0 (ODO); 1<br>(DDD-CLS) | - | Randomization group |
| gi_age | Numeric | Years | Age at enrolment |
| gi_gender | 0 (Male); 1<br>(Female) | (A) | Gender |
| hs_syncop_life | Numeric | Unit | Total number of syncope during lifetime |
| hs_syncop_lastyear | Numeric | Unit | Total number of syncope during last year |
| hs_age_syncop | Numeric | Years | Age of first syncope |
| hs_histor_presync | 0 (No); 1 (Yes) | | History of pre-syncope |
| prevepi_hosp_sync | 0 (No); 1 (Yes) | 3= | Was the patient hospitaliz ed because of syncope? |
| com_hypertension | 0 (No); 1 (Yes) | S <del>-</del> | Hypertension |
| com diabetes | 0 (No); 1 (Yes) | ide: | Diabetes |
| com_neuro_disease | 0 (No); 1 (Yes) | // <del>4</del> : | Neurological disease |
| hdis_hypertensive_disease | 0 (No); 1 (Yes) | ¥ | Hypertensive disease |
| hdis_ca_disease | 0 (No); 1 (Yes) | p= | Coronary artery disease |
| hdis_valvular_disease | 0 (No); 1 (Yes) | 1 <b>H</b> : | Valvular disease |
| hdis_hyp_cardiomyopath | 0 (No); 1 (Yes) | : <del>-</del> | Hypertrophic cardiomyopathy |
| hdis_dilated_cardiomyopath | 0 (No); 1 (Yes) | | Dilated cardiomyopathy |
| arr_fst_av_block | 0 (No); 1 (Yes) | = | First degree AV block |
| arr_atr_tachycardia | 0 (No); 1 (Yes) | De: | Atrial tachycardia |
| arr_paroxy_afib_af | 0 (No); 1 (Yes) | 14 | Paroxysmal atrial fibrillation/flutter |
| arr_perm_afib_af | 0 (No); 1 (Yes) | 5 | Permanent atrial fibrillation/flutter |
| ecg_normal_sr | 0 (No); 1 (Yes) | = | Normal sinus rhythm at enrolment |
| ecg_afib_af | 0 (No); 1 (Yes) | # | Atrial fibrillation/Flutter at enrolment |
| ecg_mean_hr | Numeric | Beats per minute | Mean heart rate |
| ecg_qrs | Numeric | msec | QRS duration |
| ecg_pr_interval | Numeric | msec | PR interval |
| echo_ejection_fraction | Numeric | % | Ejection fraction |
| ortho_supl_syst_bp | Numeric | mmHg | Supine systolic blood pressure |
| ortho_low_syst_bp | Numeric | mmHg | Lowest upright systolic blood pressure |
| ortho_max_syst_bp | Numeric | mmHg | Maximal drop in systolic blood pressure |
| carotid_rr_pause | Numeric | sec | Longest RR pause at carotid sinus massagge |
| carotid_syncope_presyncope | 0 (No); 1 (Yes) | - | Syncope or pre-syncope at carotid |



| | | | sinus massagge |
|---|---|---|---|
| cm_ace | 0 (No); 1 (Yes) | (E | ACE Inhibitors |
| cm_anticoagulant | 0 (No); 1 (Yes) | .: <del></del> | Anticoagulants |
| cm_antiplatelets | 0 (No); 1 (Yes) | 9 <del>81</del> | Antiplatelets |
| cm_b_blocker | 0 (No); 1 (Yes) | 12 | Beta-blockers |
| tt_response | 0 (Pre-syncope);<br>1 (Syncope) | | Response to tilt test |
| tt_pause_max | Numeric | sec | Maximum asystolic pause at tilt test |
| tt_pause_type | 0 (Sinus arrest);<br>1 (AV block) | * | Type of pause at tilt test |
| tt_time_pre_sync | Numeric | min | Time to symptom onset (from tilt up if positive during passive phase or from TNT administration if positive during the TNT phase) |
| tt_bp_pre_sync | Numeric | mmHg | Systolic BP at symptom onset |
| tt_low_bp | Numeric | mmHg | Lowest systolic blood pressure during tilt test |

# 7.4 Baseline data analysis

\*Baseline Analysis (STATA script)

\*Age at enrolment tabstat gi\_age, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk gi\_age ranksum gi\_age, by(rd\_display)

\*Gender tabulate gi\_gender rd\_display, chi2 column exact

\*Total number of syncope during lifetime tabstat hs\_syncop\_life, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk hs\_syncop\_life ranksum hs\_syncop\_life, by(rd\_display)

\*Total number of syncope during last year tabstat hs\_syncop\_lastyear, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk hs\_syncop\_lastyear ranksum hs\_syncop\_lastyear, by(rd\_display)

\*Age of first syncope tabstat hs\_age\_syncop, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk hs\_age\_syncop ranksum hs\_age\_syncop, by(rd\_display)

\*History of pre-syncope tabulate hs\_histor\_presync rd\_display, chi2 column exact

\*Was the patient hospitaliz ed because of syncope? tabulate prevepi\_hosp\_sync rd\_display, chi2 column exact

\*Hypertension tabulate com\_hypertension rd\_display, chi2 column exact

\*Diabetes tabulate com\_diabetes rd\_display, chi2 column exact



\*Neurological disease

tabulate com\_neuro\_disease rd\_display, chi2 column exact

\*Hypertensive disease tabulate hdis\_hypertensive\_disease rd\_display, chi2 column exact

\*Coronary artery disease tabulate hdis\_ca\_disease rd\_display, chi2 column exact

\*Valvular disease tabulate hdis\_valvular\_disease rd\_display, chi2 column exact

\*Hypertrophic cardiomyopathy tabulate hdis\_hyp\_cardiomyopath rd\_display, chi2 column exact

\*Dilated cardiomyopathy tabulate hdis\_dilated\_cardiomyopath rd\_display, chi2 column exact

\*First degree AV block tabulate arr\_fst\_av\_block rd\_display, chi2 column exact

\*Atrial tachycardia tabulate arr\_atr\_tachycardia rd\_display, chi2 column exact

\*Paroxysmal atrial fibrillation/flutter tabulate arr\_paroxy\_afib\_af rd\_display, chi2 column exact

\*Permanent atrial fibrillation/flutter tabulate arr\_perm\_afib\_af rd\_display, chi2 column exact

\*Normal sinus rhythm at enrolment tabulate ecg\_normal\_sr rd\_display, chi2 column exact

\*Atrial fibrillation/Flutter at enrolment tabulate ecg\_afib\_af rd\_display, chi2 column exact

\*Mean heart rate tabstat ecg\_mean\_hr, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk ecg\_mean\_hr ranksum ecg\_mean\_hr, by(rd\_display)

\*QRS duration tabstat ecg\_qrs, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk ecg\_qrs ranksum ecg\_qrs, by(rd\_display)

\*PR interval tabstat ecg\_pr\_interval, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk ecg\_pr\_interval ranksum ecg\_pr\_interval, by(rd\_display)

\*Ejection fraction tabstat echo\_ejection\_fraction, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk echo\_ejection\_fraction ranksum echo\_ejection\_fraction, by(rd\_display)

\*Supine systolic blood pressure tabstat ortho\_supl\_syst\_bp, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk ortho\_supl\_syst\_bp ranksum ortho\_supl\_syst\_bp, by(rd\_display)

\*Lowest upright systolic blood pressure tabstat ortho\_low\_syst\_bp, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics)



swilk ortho\_low\_syst\_bp
ranksum ortho\_low\_syst\_bp, by(rd\_display)

\*Maximal drop in systolic blood pressure tabstat ortho\_max\_syst\_bp, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk ortho\_max\_syst\_bp ranksum ortho\_max\_syst\_bp, by(rd\_display)

\*Longest RR pause at carotid sinus massagge tabstat carotid\_rr\_pause, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk carotid\_rr\_pause ranksum carotid\_rr\_pause, by(rd\_display)

\*Syncope or pre-syncope at carotid sinus massagge tabulate carotid\_syncope\_presyncope rd\_display, chi2 column exact

\*ACE Inhibitors tabulate cm\_ace rd\_display, chi2 column exact

\*Anticoagulants tabulate cm\_anticoagulant rd\_display, chi2 column exact

\*Antiplatelets tabulate cm\_antiplatelets rd\_display, chi2 column exact

\*Beta-blockers tabulate cm\_b\_blocker rd\_display, chi2 column exact

\*Response to tilt test tabulate tt\_response rd\_display, chi2 column exact

\*Maximum asystolic pause at tilt test tabstat tt\_pause\_max, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk tt\_pause\_max ranksum tt\_pause\_max, by(rd\_display)

\*Type of pause at tilt test tabulate tt\_pause\_type rd\_display, chi2 column exact

\*Time to symptom onset(from tilt up if positive during passive
\*phase or from TNT administration if positive during the TNT phase)
tabstat tt\_time\_pre\_sync, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics)
swilk tt\_time\_pre\_sync
ranksum tt\_time\_pre\_sync, by(rd\_display)

\*Systolic BP at symptom onset tabstat tt\_bp\_pre\_sync, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk tt\_bp\_pre\_sync ranksum tt\_bp\_pre\_sync, by(rd\_display)

\*Lowest systolic blood pressure during tilt test tabstat tt\_low\_bp, statistics(mean sd p50 p75 p25) by(rd\_display) columns (statistics) swilk tt\_low\_bp ranksum tt\_low\_bp, by(rd\_display)





# 7.5 Evaluation of study objectives

The BIOSync CLS study (BA103, CIP ver. 7.0) gathers primary and secondary endpoints' data through self-administered patient questionnaires. In order to ensure double-blinding in endpoint assessment, the questionnaires will be collected by external personnel of an appointed CRO. This process is descripted in detail in the Charter for patient questionnaire collection and adjudication, version 2.0, 06-Mar-2017, and summarized in the below image.



At the end of the adjudication the following derived variables will be created.

| Variable name | List of values | Unit of measure | Description |
|---|---|---|---|
| pe | 0 (No); 1 (Yes) | * | Occurrence of syncope episode |
| time_pe | Numeric | days | If pe=1: time to the first post |
| | | | randomization recurrence of a |
| | | | syncopal episode; |
| | | | If pe=0: total follow-up time |
| se | 0 (No); 1 (Yes) | - | Occurrence of pre-syncope or |
| | | | syncope episode |
| time_pe | Numeric | days | If pe=1: time to the first post |
| | | | randomization recurrence of a pre- |
| | | | syncope or syncope episode |
| | | | whichever comes first.; |
| | | | If pe=0: total follow-up time |

The analysis of the primary and secondary study objectives will be performed with the following code (STATA language).

stset time\_pe, failure(pe==1)

\*Kaplan\_meier plots generation

sts graph by(rd\_display), ci risktable

\*Comparison of survivors functions

sts test rd\_display, logrank

\*Proportional hazard Cox models for major baseline predictors

stcox rd display

estat phtest

stcox gi\_age

stcox gi\_gender

stcox hs syncop life

stcox hs\_syncop\_lastyear

stcox ecg\_mean\_hr

stcox tt\_response

stcox tt\_pause\_max

stcox tt\_pause\_type

stcox tt\_time\_pre\_sync



<sup>\*</sup>Study objectives evaluation

<sup>\*</sup>Primary endpoint

\*Secondary endpoint

stset time\_se, failure(se==1)

\*Kaplan\_meier plots generation
sts graph, by(rd\_display) ci

\*Comparison of survivors functions
sts test rd\_display, logrank

\*Proportional hazard Cox models for major baseline predictors
stcox rd\_display
estat phtest
stcox gi\_age
stcox gi\_gender

stcox hs\_syncop\_lastyear stcox ecg\_mean\_hr

stcox tt\_response stcox tt\_pause\_max

stcox hs\_syncop\_life

stcox tt\_pause\_type stcox tt\_time\_pre\_sync

stcox tt\_low\_bp

# 7.6 Interim analysis

Interim analyses will be performed at t=0.4 and 0.7 of the required primary endpoint events or, equivalently, after 25 and 43 endpoint events will be collected. The final analysis will be performed after the study database has been closed out. In order to keep the overall type I error at the level of 0.05, two-sided, symmetric O'Brien-Fleming boundaries generated with the Lan-DeMets spending function approach to group-sequential testing will be assumed as early stopping rules for efficacy.

| t | 0.40 | 0.70 | 1.00 |
|---------------------|---------|---------|---------|
| No. endpoint events | 25 | 43 | 62 |
| Zup | 3.3569 | 2.4445 | 2.0005 |
| $Z_{low}$ | -3.3569 | -2.4445 | -2.0005 |
| р | 0.0008 | 0.015 | 0.05 |

# 7.7 Clinical Investigation Plan (CIP) deviations

All CIP deviations will be classified with details of the type of deviation and the full-list will be provided in the Clinical Investigational Report (CIR).

The number (and percentage) of patients with major and minor protocol deviations will be summarized by randomization group.

A post-hoc per-protocol analysis according to the existing data gathered could be run after the evaluation of the provided deviations.



Page 14/14

### References

- (1) Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martín A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018; 39(21):1883-1948.
- (2) Brignole M, Menozzi C, Moya A, Andresen D, Blanc JJ, Krahn AD, Wieling W, Beiras X, Deharo JC, Russo V, Tomaino M, Sutton R; International Study on Syncope of Uncertain Etiology 3 (ISSUE-3) Investigators. Pacemaker therapy in patients with neurally mediated syncope and documented asystole: Third International Study on Syncope of Uncertain Etiology (ISSUE-3): a randomized trial. Circulation. 2012; 125(21): 2566-71.

